CLINICAL TRIAL: NCT05378724
Title: Effectiveness of Hospital Fit on Physical Activity of Hospitalised Patients: a Stepped-wedge Cluster-randomised Clinical Trial and Process Evaluation
Brief Title: Effectiveness of Hospital Fit on Physical Activity of Hospitalised Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NL
Record Dates: First submitted 2022-04-08; First posted 2022-05-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2022-09

CONDITIONS: Cardiovascular Diseases; Oncology; Activation, Patient
Keywords: Physical activity; eHealth; Accelerometer; Hospitalization; Effectiveness; Process evaluation
MeSH Terms: conditions — Cardiovascular Diseases; Neoplasms; Patient Participation; Motor Activity

STUDY DESIGN:
Intervention Model Description: A prospective, multi-center, stepped-wedge cluster-randomised trial will be performed to investigate the effectiveness of Hospital Fit. Additionally, a process evaluation will be performed using semi-structured interviews and questionnaires in patients and focus-group interviews in healthcare professionals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): All subjects eligible for inclusion in this study will receive usual care physiotherapy treatment. The number of treatment sessions and content of physiotherapy treatment sessions will depend on the diagnosis and needs of the individual patient. This study will not interfere with the content of the usual care physiotherapy treatment. Usual care physiotherapy sessions wil take approximately 20-30 minutes per session. They receive no additional intervention and will not use Hospital Fit as part of their physiotherapy treatment. The patients in the control group will receive an activity monitor to collect data about their physical activity levels. However, patients and their healthcare professionals will not receive feedback on patients' physical activity levels.
- Intervention group (Experimental): Patients in the intervention group will receive usual care physiotherapy and us Hospital Fit additionally. At the end of the last physiotherapy treatment session before discharge, or after a maximum of nine days of study inclusion (whichever comes first), the physiotherapist will remove the activity monitor and data collection will end.
  Interventions: Device: Hospital Fit 2.0, HFITAPP0, release 05, Maastricht Instruments B.V., the Netherlands

INTERVENTIONS:
Device: Hospital Fit 2.0, HFITAPP0, release 05, Maastricht Instruments B.V., the Netherlands — Hospital Fit consists of a smartphone app combined to the MOX accelerometer. Hospital Fit provides patients and physiotherapists direct feedback on patients' physical activity behavior. Individual goals regarding the number of minutes per day spent walking can be set by the therapist. Hospital Fit also gives patients insight into their own recovery process. During every treament, the physiotherapist will evaluate the extent of functional recovery. In addition, Hospital Fit will give physiotherapists the option of creating a patient-specific exercise program supported by videos. During every treatment session, the patient and physiotherapist will evaluate (and if necessary adapt) the amount of activity performed since the previous treatment, the extent of functional recovery and the exercise program.
  Arms: Intervention group

SUMMARY:
The primary objective of this study is to investigate the effectiveness of using Hospital Fit as part of the physiotherapy treatment on average time spent walking per day in patients hospitalised at the Medical Oncology or Cardiology Departments of the Maastricht University Medical Center (MUMC+) and Radboud University Medical Center (Radboudumc) compared to patients who received physiotherapy before implementation of Hospital Fit. Secondary: to investigate the effectiveness of using Hospital Fit as part of the physiotherapy treatment on average time spent standing per day, average time spent lying/sitting per day, average number of transitions per day and the Modified Iowa Level of Assistance scale (mILAS) scores in hospitalised patients. Besides, the reach, efficacy, adoption, and implementation of using Hospital Fit as part of the physiotherapy treatment will be investigated from the perspective of both patients and healthcare professionals.

DETAILED DESCRIPTION:
Rationale: Physical inactivity is a major, underrecognised problem in patients during their hospital stay. Patients spend between 87 and 100% of their time lying or sitting. This physical inactivity has been associated with adverse outcomes such as functional decline, increased length of hospital stay and mortality. Digital health tools could be valuable to prevent negative effects of inactivity. Hospital Fit is a promising app-based intervention to stimulate physical activity by 1) continuous physical activity monitoring, 2) personalised goalsetting, 3) providing patients insight in their functional recovery, 4) providing patients tailored exercise programs, 5) informing patients about benefits of physical activity, and 6) reminding patients to use Hospital Fit 7) linking the data to the electronic medical record, making it available for other healthcare professionals.

Objectives: Primary: to investigate the effectiveness of using Hospital Fit as part of the physiotherapy treatment on average time spent walking per day in patients hospitalised at the Medical Oncology or Cardiology Departments of the Maastricht University Medical Center (MUMC+) and Radboud University Medical Center (Radboudumc) compared to patients who received physiotherapy before implementation of Hospital Fit. Secondary: 1) to investigate the effectiveness of using Hospital Fit as part of the physiotherapy treatment on average time spent standing per day, average time spent lying/sitting per day, average number of transitions per day and the Modified Iowa Level of Assistance scale (mILAS) scores in hospitalised patients; and 2) to investigate the reach, efficacy, adoption, and implementation of using Hospital Fit as part of the physiotherapy treatment from the perspective of both patients and healthcare professionals.

Study design: A prospective, multi-centre, stepped-wedge cluster randomised trial will be performed to investigate the effectiveness of Hospital Fit. Additionally a process evaluation will be performed using questionnaires and semi-structured interviews in patients and focus-group interviews in healthcare professionals.

Study population: In total 180 patients hospitalised at the Medical Oncology Department or Cardiology Departments at the MUMC+ or Radboudumc will be included to study the effectiveness. The process evaluation will be performed in the intervention group using a questionnaire in all 90 patients, semi-structured interviews in 24 purposefully selected patients (or less if data saturation is reached), and focus group interviews in 24 healthcare professionals (i.e., physiotherapists, nurses, and physicians (assistants).

Intervention: Physical activity will be measured in all patients with an accelerometer until discharge with a maximum of nine days. The control group will receive usual care physiotherapy (n=90), while the intervention group will use Hospital Fit additionally (n=90).

Main study parameters/endpoints: Primary outcome parameter: average time spent walking per day (min). Secondary outcome parameters: average time spent standing and lying/sitting per day (min.), average number of transitions from lying/sitting to standing/walking per day, and mILAS score per day. Outcome parameters process evaluation: participation; representation; perceived efficacy; use of app; use of different functionalities; barriers and facilitators to Hospital Fit use; and expected maintenance.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The burden and risks on patients are minimal. The control group will receive usual care physiotherapy and will wear an accelerometer. The intervention group will use Hospital Fit additionally. Wearing a small accelerometer and using Hospital Fit should not be a burden to patients. The only burden is the time it takes to prepare subjects (install app, explain study). No invasive interventions will take place. Anticipated benefits of Hospital Fit use include improved physical activity, therewith reducing the negative effects associated with low physical activity.

ELIGIBILITY:
Inclusion Criteria patients:

* Over 18 years old.
* Receiving physiotherapy at the Medical Oncology Department or the Cardiology Department at the MUMC+ or Radboudumc.
* Enough understanding of the Dutch language.
* Owning a smartphone (operating system: at least iOS 13.0 or Android 8.0).
* Able to use a smartphone app.
* Able to walk independently 2 weeks before admission, as scored on the Functional Ambulation Categories (FAC >3).

Exclusion Criteria patients:

* A contraindication to walking (as reported by a medical specialist in the electronic medical record).
* A contraindication to wearing an activity monitor, fixed by a hypoallergenic plaster at the upper leg (such as active bilateral upper leg infection, severe oedema or bilateral transfemoral amputation).
* Admitted for cancers of the head and neck (i.e., cancer in the oral cavity, throat (pharynx), voice box (larynx), paranasal sinuses and nasal cavity, salivary glands).
* Admitted with cardiac arrhythmia and hemodynamic instability requiring medication over 48 hours (i.e., beta blockers or noradrenaline) or invasive treatment (i.e., pacemaker or defibrillator implementation).
* Mentally incapacitated subjects as reported by healthcare professionals in the medical record. When any doubt arises, the patient will be excluded.
* Impaired cognition (delirium / dementia) as reported in the medical record by a healthcare professional. When any doubt arises, the patient will be excluded.
* Unable to participate in the informed consent procedure or unable to provide written informed consent.
* A life expectancy shorter than 3 months as mentioned by the medical specialist in the medical record.
* Previous participation in this study.

Inclusion Criteria healthcare professionals:

* Employed as physiotherapist, nurse or physician (assistant) at the Medical Oncology Department or the Cardiology Department.
* Working at the MUMC+ or Radboudumc for at least one month.

Exclusion Criteria healthcare professionals:

• No participation in care for patients at the Medical oncology Department or Cardiology Department during the intervention phase (e.g., absence or research employment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Average time spent walking per day (minutes). | Period between inclusion and discharge, with a maximum of nine days.
  Total number of minutes walking divided by the total number of valid measurement days in the period between inclusion and discharge, with a maximum of nine days.

SECONDARY OUTCOMES:
Average time spent standing per day (minutes). | Period between inclusion and discharge, with a maximum of nine days.
  Total number of minutes standing divided by the total number of valid measurement days in the period between inclusion and discharge, with a maximum of nine days.
Average time spent lying/sitting per day (minutes). | Period between inclusion and discharge, with a maximum of nine days.
  Total number of minutes lying/sitting divided by the total number of valid measurement days in the period between inclusion and discharge, with a maximum of nine days.
Average number of transitions per day from a sedentary position (lying or sitting) to an active position (standing or walking). | Period between inclusion and discharge, with a maximum of nine days.
  Total number of transitions divided by the total number of valid measurement days in the period between inclusion and discharge, with a maximum of nine days.
Modified Iowa Level of Assistance scale (mILAS) scores per day. | Period between inclusion and discharge, with a maximum of nine days.
  The 5-item Modified Lowa Level of Assistance Scale (mILAS) assesses the ability of patients to perform 5 activities of daily living and rates the amount of assistance and type of walking aid needed. Each item has a 7-point rating scale (0-6 points), resulting in total scores ranging between 0-30 points. Higher scores indicate that a patient needs more assistance.

OTHER OUTCOMES:
Reach - Participation: Percentage of users (patients) of Hospital Fit that is reached in the intervention phase | Period between inclusion and discharge with a maximum of nine days
  The 'total number of users' (included patients allocated to the intervention group that used Hospital Fit) divided by the 'total number of included subjects' (all included patients allocated to the intervention group). A 'user' is defined included subject who has indicated that she/he used Hospital Fit at least once.
Reach - Representation: Patient characteristics of users and non-users in | Period between inclusion and discharge with a maximum of nine days
  Patient characteristics (i.e., age, gender, clinical diagnosis) of patients in the intervention group shown separate for users and non-users. A 'user' is defined included subject who has indicated that she/he used Hospital Fit at least once. A 'non-user' is an included subject who has indicated in the questionnaire that she/he did not use Hospital Fit.
Efficacy - Perceived efficacy | Patient interviews at day of removal of accelerometer (=day of discharge or after max. 9 days of Hospital Fit use (whichever comes first)). Healthcareprofessional interviews: after the last patient has terminated the study (Jan.2023).
  Data on perceived efficacy will be collected using individual, semi-structured, face-to-face interviews with 24 patients included in the intervention group and 4 focus group interviews with in total 6 healthcare professionals (physiotherapists, nurses, and physician(s) assistant(s)) per focus group. The following topics will be discussed: What is the impact of Hospital Fit use on physical activity of patients during their hospital stay according to patients? How do healthcare professionals determine if Hospital Fit use has been effective for patients? What were perceived positive and negative outcomes? How likely is it that Hospital Fit improved patients' physical activity?
Adoption - Use of app: Frequency of Hospital Fit use per day | Period between inclusion and discharge, with a maximum of nine days
  Patients included in the intervention roup will score how many times per day she/he has used Hospital Fit on a daily questionnaire.
Adoption - Use of different functionalities per day: Use of different functionalities of Hospital Fit | Period between inclusion and discharge, with a maximum of nine days
  Patients included in the intervention group will score how many times per day the different functionalities of Hospital Fit were used on a daily questionnaire.
Implementation - Barriers and facilitators to Hospital Fit use | Patient interviews at day of removal of accelerometer (=day of discharge or after max. 9 days of Hospital Fit use (whichever comes first)). Healthcareprofessional interviews: after the last patient has terminated the study (Jan.2023)
  Barriers and facilitators to Hospital Fit use according to patients allocated to the intervention group and healthcare professionals. This will be explored using individual, semi-structured, face-to-face interviews with 24 patients included in the intervention group and 4 focus group interviews with in total 6 healthcare professionals (physiotherapists, nurses, and physician(s) assistant(s)) per focus group.
Maintenance - Expected maintenance | Patient interviews at day of removal of accelerometer (=day of discharge or after max. 9 days of Hospital Fit use (whichever comes first)). Healthcareprofessional interviews: after the last patient has terminated the study (Jan.2023)
  Expected maintenance will be explored using individual, semi-structured, face-to-face interviews with 24 patients included in the intervention group and 4 focus group interviews with in total 6 healthcare professionals (physiotherapists, nurses, and physician(s) assistant(s)) per focus group. The following topics will be discussed: What might be the long-lasting effects of Hospital Fit on physical activity of patients? How will Hospital Fit be maintained at the hospital ward?

CONTACTS AND LOCATIONS:
Overall Officials: Antoine F Lenssen, Prof, PhD, Principal Investigator — Maastricht University Medical Center
Locations (2):
- Netherlands (2):
  - Radboudumc, Nijmegen, Gelderland
  - MaastrichtUMC, Maastricht, Limburg

IPD SHARING:
Plan to Share IPD: No
We do not intent to make IPD available to other researchers.